CLINICAL TRIAL: NCT03332836
Title: A Phase 1, Multiple Ascending Dose, Glucose Clamp Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HM12460A Compared to Insulin Glargine in Subjects With Type 2 Diabetes Mellitus
Brief Title: Multiple Ascending Dose Study of HM12460A in Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sopnsor decision
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-INS-102
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single dose subcutaneous administration (Dose A)
  Interventions: Biological: HM12460A
- Cohort 2 (Experimental): Single dose subcutaneous administration (Dose B)
  Interventions: Biological: HM12460A
- Cohort 3 (Experimental): Single dose subcutaneous administration (Dose C)
  Interventions: Biological: HM12460A

INTERVENTIONS:
Biological: HM12460A — HM12460A is a long-acting insulin

SUMMARY:
This is a phase 1 multiple ascending dose (MAD) study, conducted in subjects with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Female subjects must be non-pregnant and non-lactating

Exclusion Criteria:

* Recurrent severe hypoglycemia or hypoglycemic unawareness or recent severe ketoacidosis, as judged by the Investigator
* Pregnant or lactating women
* Participation in an investigational study within 30 days prior to dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 month
  An adverse event is any undesirable and unintended medical event occurring to a subject in a clinical study, whether or not related to the investigational products.

SECONDARY OUTCOMES:
Cmax of HM12460A | 1 month
  - Maximum concentration of HM12460A over the entire dosing period
AUC of HM12460A | 1 month
  - Area Under the Curve of HM12460A over the entire dosing period

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Investigative Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided